CLINICAL TRIAL: NCT04215042
Title: Prevention of Contrast-Induced Acute Kidney Injury: Standard Versus Short Hydration Protocol in Patients With Normal Fluid Status Assessed by the Bioimpedance Analysis (The HYDRA II Study)
Brief Title: Tailored Hydration Based on Bioimpedance Analysis for Prevention of Contrast Induced Acute Kidney Injury
Acronym: Hydra2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Misericordia e Dolce (Other)
Responsible Party: Principal Investigator, Mauro Maioli, Medical Doctor - Cardiology, Ospedale Misericordia e Dolce
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Prato0707
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Acute Kidney Injury
Keywords: Contrast-Induced Acute Kidney Injury; Contrast-Induced Nephropathy; Contrast-Associated Acute Kidney Injury; Contrast media; Angiography; Coronary percutaneous intervention
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard hydration (Active Comparator): All patients received standard intravenous saline hydration (0.9% sodium chloride, 1 ml/kg/h for 12 hours before and 6 hours after procedure
  Interventions: Drug: sodium chloride infusion
- Short hydration (Experimental): All patients received shot intravenous saline hydration (3 ml/kg for 1 hour before the procedure and after 1ml/kg/h for 6 hours)
  Interventions: Drug: sodium chloride infusion

INTERVENTIONS:
Drug: sodium chloride infusion

SUMMARY:
The aim of this study was to evaluate, in patients with "normal fluid status" assessed by the bio-impedance analysis, whether two different protocol of IV isotonic saline infusion are associated with different volume expansion and differing risks for Contrast Induced Acute Kidney Injury in patients undergoing coronary angiographic procedure.

DETAILED DESCRIPTION:
Iodinated contrast media are a well-recognized cause of iatrogenic acute kidney injury in patients undergoing imaging diagnostic or therapeutic procedures (contrast-induced acute kidney injury, CI-AKI). Extracellular volume expansion at the time of contrast media administration may represent important protective strategies that play a major role in the prevention CI-AKI.

Bio-impedance analysis is an inexpensive, rapid, and accurate tool for evaluating a patient's hydration status, and can be performed at the bedside within minutes [Maioli, Journal of American College Cardiology 1014;63:1387-94]. In this study we defined patients with "lower fluid status" with high risk of CI-AKI (Male with resistance/ height ratio > 315 Ohm/meter and Female > 380 Ohm/meter). Bio-impedance analysis IVA may represent the optimal tool to monitor the adequacy of volume expansion and protective strategy delivery.

Infusing a standardized amount of fluid before the procedure may not result in the same effects in all patients. Moreover, standardized fluid infusion for 24 hours in patients that present with "normal fluid status" assessed by the bioimpedance analysis, can represent a too expensive preventive option both in terms of care and discomfort for the patient. In this study we analyze the possibility of a non-inferiority preventive protocol that involves a lower infusion of saline solution with a shorter administration time.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients admitted in Cardiology Unit for coronary or peripheral angiography with "normal fluid status" assessed on the basis bio-impedance analysis (Male with resistance/height ratio < 315 Ohm/meter and female < 380 Ohm/meter)

Exclusion Criteria:

* contrast medium administration within the 10 days
* end stage renal failure requiring dialysis
* no ability to evaluation the state of hydration with bio impedance
* refused to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of contrast induced acute kidney injury (CI-AKI) | 1 day
  CI-AKI is defined as an increase in serum Cystatin C concentration 10%, above the baseline value, at 24 hours after administration of contrast medium

SECONDARY OUTCOMES:
incidence of contrast induced acute kidney injury (CI-AKI) | 2 days
  CI-AKI is defined as an increase in serum Creatinine >= 0,3 mg/dL over baseline value within 2 days after the administration of contrast medium

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Santo Stefano, Prato, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maioli M, Toso A, Leoncini M, Musilli N, Bellandi F, Rosner MH, McCullough PA, Ronco C. Pre-procedural bioimpedance vectorial analysis of fluid status and prediction of contrast-induced acute kidney injury. J Am Coll Cardiol. 2014 Apr 15;63(14):1387-94. doi: 10.1016/j.jacc.2014.01.025. Epub 2014 Feb 12. PMID 24530668
- [Background] Maioli M, Toso A, Leoncini M, Musilli N, Grippo G, Ronco C, McCullough PA, Bellandi F. Bioimpedance-Guided Hydration for the Prevention of Contrast-Induced Kidney Injury: The HYDRA Study. J Am Coll Cardiol. 2018 Jun 26;71(25):2880-2889. doi: 10.1016/j.jacc.2018.04.022. PMID 29929610